CLINICAL TRIAL: NCT01960972
Title: Launching a Salt Substitute to Reduce Blood Pressure at the Population Level - Peru
Brief Title: Launching a Salt Substitute to Reduce Blood Pressure at the Population Level in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jaime Miranda, Research Professor, Universidad Peruana Cayetano Heredia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5U01HL114180 (NIH); 58563 (Other: UPCH SIDISI); 00004928 (Other: JHU IRB)
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Blood Pressure; Hypertension
Keywords: Blood pressure; Hypertension; Stepped wedge trial design
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salt substitute (Experimental): As described by Brown, in a stepped wedge design, an intervention is rolled-out sequentially to the trial participants (either as individuals or clusters of individuals) over a number of time periods. The order in which the different individuals or clusters receive the intervention is determined at random and, by the end of the random allocation, all individuals or groups will have received the intervention. Stepped wedge designs incorporate data collection at each point where a new group (step) receives the intervention.
  Thus, the salt substitute will be implemented in each cluster (village) in a randomized fashion. Not arms are needed since the 6 randomly-selected villages will be implemented in some moment of the protocol.
  Interventions: Other: Salt substitute

INTERVENTIONS:
Other: Salt substitute — A salt substitute using 25% of potassium chloride and 75% of sodium chloride will be implemented in each of the villages.

SUMMARY:
This protocol aims to implement, using a stepped wedge trial design, a population-level intervention to replace high-sodium salt for a salt substitute (low-sodium, high-potassium salt) to reduce blood pressure levels among adults aged 18 years and over of the semi-urban area of Tumbes.

We hypothesize that participants aged 18 years and over from villages receiving a salt substitute will have lower blood pressure compared to control villages.

DETAILED DESCRIPTION:
Several randomized clinical trials and meta-analysis have reported that reduction of sodium intake decreases blood pressure. Also, the increase of potassium ingestion in minimal doses has been found in systematic reviews to produce a small reduction in blood pressure levels.

The proposed intervention is a community-wide mass-strategy in which direct delivery of a salt substitute to households is accompanied by wide social marketing campaigns, both before and during the intervention period. With this experimental stepped wedge trial design, we will estimate the impact of a reduced-sodium salt substitution program on blood pressure at the population level.

We propose the following specific aims:

Specific Aim 1: To implement and assess the impact of an intervention using a salt substitute on blood pressure at the population level using a stepped wedge trial design.

Specific Aim 2: To determine costs and efficacy of this implementation strategy using cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years and over from the randomly selected villages.
* Capable of understanding study procedures and providing informed consent.
* Full-time resident in the area.

Exclusion Criteria:

* Self-reported history of chronic kidney disease or heart disease.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2376 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Systolic/diastolic blood pressure (mmHg) | Three years
  We will assess changes in systolic and diastolic blood pressure over time. Periodic assessments will be carried out to obtain clinical measurements. Every five months, a new evaluation will be performed in all participant villages (intervention and control).
  Systolic and diastolic blood pressure will be measured in triplicate using standard procedures and automated and validated devices. These periodic assessments will be taken at each household to guarantee contact with each family member enrolled in this study.

SECONDARY OUTCOMES:
Progression to hypertension | Three years
  Using data of systolic and diastolic blood pressure, we will estimate progression towards hypertension among participants in intervened and control villages.

OTHER OUTCOMES:
Cost-effectiveness analysis | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Miranda, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Robert H Gilman, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Antonio Bernabe-Ortiz, MD, MPH, Study Director — Universidad Peruana Cayetano Heredia
Locations (1):
- Center for Global Health (Universidad Peruana Cayetano Heredia), Tumbes, Peru

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared potentially when main papers are published.

REFERENCES:
- [Background] Bernabe-Ortiz A, Diez-Canseco F, Gilman RH, Cardenas MK, Sacksteder KA, Miranda JJ. Launching a salt substitute to reduce blood pressure at the population level: a cluster randomized stepped wedge trial in Peru. Trials. 2014 Mar 25;15:93. doi: 10.1186/1745-6215-15-93. PMID 24667035
- [Result] Pesantes MA, Diez-Canseco F, Bernabe-Ortiz A, Ponce-Lucero V, Miranda JJ. Taste, Salt Consumption, and Local Explanations around Hypertension in a Rural Population in Northern Peru. Nutrients. 2017 Jul 5;9(7):698. doi: 10.3390/nu9070698. PMID 28678190
- [Result] Saavedra-Garcia L, Bernabe-Ortiz A, Gilman RH, Diez-Canseco F, Cardenas MK, Sacksteder KA, Miranda JJ. Applying the Triangle Taste Test to Assess Differences between Low Sodium Salts and Common Salt: Evidence from Peru. PLoS One. 2015 Jul 30;10(7):e0134700. doi: 10.1371/journal.pone.0134700. eCollection 2015. PMID 26225848
- [Result] Bernabe-Ortiz A, Sal Y Rosas VG, Ponce-Lucero V, Cardenas MK, Carrillo-Larco RM, Diez-Canseco F, Pesantes MA, Sacksteder KA, Gilman RH, Miranda JJ. Effect of salt substitution on community-wide blood pressure and hypertension incidence. Nat Med. 2020 Mar;26(3):374-378. doi: 10.1038/s41591-020-0754-2. Epub 2020 Feb 17. PMID 32066973
- [Derived] Lazo-Porras M, Del Valle A, Beran D, Pesantes MA, Perez-Leon S, Ponce-Lucero V, Bernabe-Ortiz A, Cardenas MK, Chappuis F, Perel P, Miranda JJ, Diez-Canseco F. Implementation of a salt substitute intervention using social marketing in resourced-limited communities in Peru: a process evaluation study. Front Public Health. 2023 May 19;11:1068624. doi: 10.3389/fpubh.2023.1068624. eCollection 2023. PMID 37275501